CLINICAL TRIAL: NCT00233012
Title: A Randomized, Open-label (OL), Multicenter Study With OL Extension of the Pharmacokinetics and Safety of Topiramate Administered as Oral Liquid and Sprinkle Formulations as an Adjunct to Concurrent Anticonvulsant Therapy in Infants (Aged 1-24 Months, Inclusive) With Refractory Partial-onset Seizures
Brief Title: A Study of the Pharmacokinetics, Safety and Tolerability of Topiramate in Infants (Age 1-24 Months) With Refractory Partial-onset Seizures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Other Study IDs: CR002236
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Seizures
Keywords: Refractory partial-onset seizures; Infants aged 1-24 months; Pharmacokinetics; Topiramate
MeSH Terms: conditions — Seizures | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics safety and tolerability of topiramate in infants aged 1-24 months with refractory partial-onset seizures. Topiramate is an antiepileptic drug approved for use in adult and pediatric patients (aged 2 to 16 years) with refractory partial onset seizures (POS) with or without secondarily generalized seizures, primary generalized tonic clonic seizures, or Lennox-Gastaut syndrome (LGS).

DETAILED DESCRIPTION:
This is a open-label, randomized (patients are assigned different treatments based on chance), dose comparison, multicenter study of topiramate in infants of age 1-24 months with refractory partial-onset seizures (POS). The trial will evaluate the pharmacokinetics, safety, and tolerability of topiramate used as additional treatment in infants with refractory POS. Topiramate is administered as liquid and sprinkles as adjunct (additional treatment) to concurrent anticonvulsant therapy. The study will consist of 4 phases: a pretreatment phase that includes screening (up to 7 days) and baseline (1 day), an open-label treatment phase (up to 6 weeks), an open-label extension phase (54 weeks), and a posttreatment phase (up to 4 weeks). Seizure diaries will be maintained throughout the study by the patients' parents, legally acceptable representatives, or caregivers. In the open-label treatment phase, patients will be randomly assigned to 1 of 4 treatments: topiramate 3, 5, 15, or 25 mg/kg per day. Venous blood samples (four 1 milliliter [mL] samples) will be collected on 2 days during the study to determine plasma concentration of topiramate. Safety will be evaluated throughout the study by monitoring adverse events and by results from clinical laboratory tests (serum chemistry, venous ammonia, hematology, and urinalysis), electrocardiograms (ECGs), vital sign measurements (pulse and blood pressure), physical examination, neurologic examination, Vineland Scales of Adaptive Behavior, renal ultrasound, assessments for adequate food and liquid intake, hyperthermia, oligohydrosis, and rash, and take-home records. Liquid or sprinkles form of topiramate, 3,5,15,or 25mg/kg per day for 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Regular enteral feeding (solid food
* bottle- or cup-fed) with or without breastfeeding
* weigh >/=3.5 kilograms (kg) and <15.5 kg
* Length using an infant measuring table (heel to crown) must be = 49 cm
* clinical or electroencephalographic (EEG) evidence of POS (simple or complex) with or without secondary generalization of at least 1 month in duration in infants >6 months of age, or at least 2 weeks in duration in infants <6 months of age
* Multiple seizure types allowed as long as POS is present
* Taking 1 or 2 concurrent marketed antiepileptic drugs (AEDs) for >1 month for infants >6 months of age and for >2 weeks for infants <6 months of age
* the regimen of AEDs at entry must be considered inadequate in controlling seizures, after being optimized in the opinion of the investigator
* Have had a computerized tomography or magnetic resonance imaging scan to confirm the absence of a progressive lesion such as a tumor, with the exception of lesions of tuberous sclerosis and Sturge-Weber syndrome, which are allowed.

Exclusion Criteria:

* Exclusively breast-fed and cannot take oral liquid medication
* Receives regular enteral feeding using gastrostomy, jejunostomy, or nasogastric tube
* have surgically implanted and functioning vagus nerve stimulator
* Have febrile seizures or seizures due to an acute medical illness
* Have infantile seizures as a result of a correctable medical condition such as metabolic disturbance, toxic exposure, neoplasm, or active infection
* History of nonepileptic seizures, either current or at any point in the past
* Any progressive neurologic disorder, including malignancy, brain tumor, active central nervous system infection, demyelinating disease, or degenerative or progressive central nervous system disease with the exception of tuberous sclerosis and Sturge Weber syndrome.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2005-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Individual (each patient) and mean (each treatment) topiramate plasma concentration-time profiles.

SECONDARY OUTCOMES:
Incidence of adverse events throughout the study. Changes from pretreatment to the end of posttreatment phase in take-home records, clinical laboratory results, physical & neurologic examination results, ECGs, renal ultrasounds, vital sign measurements

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Ness S, Todd MJ, Wang S, Eerdekens M, Nye JS, Ford L. Adaptive behavior outcomes in infants treated with adjunctive topiramate. Pediatr Neurol. 2012 Jun;46(6):350-8. doi: 10.1016/j.pediatrneurol.2012.02.028. PMID 22633629
- [Derived] Puri V, Ness S, Sattaluri SJ, Wang S, Todd M, Yuen E, Eerdekens M, Nye JS, Manitpisitkul P, Shalayda K, Ford L. Long-term open-label study of adjunctive topiramate in infants with refractory partial-onset seizures. J Child Neurol. 2011 Oct;26(10):1271-83. doi: 10.1177/0883073811406982. Epub 2011 Jun 14. PMID 21673279